CLINICAL TRIAL: NCT05306106
Title: Determination of the Glycemic Index of Pastry. A Randomized Study on Healthy Volunteers.
Brief Title: Glycemic Index of Pastry
Acronym: IG-DESSERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, Principal investigator, Institut Pasteur de Lille
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2020-A03161-38
Record Dates: First submitted 2021-10-11; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: pastry; glycemic index
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Intervention Model Description: monocentric, randomized, cross-over and ambulatory study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Glucose (Other): The control product, said to be the reference product, is an oral solution of 50 g of glucose.
  Interventions: Other: Glucose
- a truffle match (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: truffle match
- a hazelnut chocolate cookie (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: hazelnut chocolate cookie
- a Paris Brest style eclair (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: Paris Brest style eclair
- a hazelnut chocolate finger (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: hazelnut chocolate finger
- a lemon finger (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: lemon finger
- a elderflower madeleine (Other): The products evaluated are pastries from the Mademoiselle Desserts range, namely a truffle match, a hazelnut chocolate cookie, a Paris Brest style eclair, a hazelnut chocolate finger, a lemon finger and an elderflower madeleine.
  Interventions: Other: elderflower madeleine

INTERVENTIONS:
Other: Glucose — Each subject will consume the reference product during visits V1 and V5. A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume the glucose solution. The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: Glucose
Other: truffle match — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 221.2 g of truffle match (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a truffle match
Other: hazelnut chocolate cookie — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 142.8 g of hazelnut chocolate cookie (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a hazelnut chocolate cookie
Other: Paris Brest style eclair — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 277.7 g of Paris Brest style eclair (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a Paris Brest style eclair
Other: hazelnut chocolate finger — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 312.5 g of hazelnut chocolate finger (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a hazelnut chocolate finger
Other: lemon finger — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 263.1 g of lemon finger (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a lemon finger
Other: elderflower madeleine — The products evaluated are pastries from the Mademoiselle Desserts range. The amounts consumed will be calculated for each of the pastries so that 50 g of carbohydrate is ingested per intake. Subjects may consume 200 mL of water after ingesting the pastries. During visits V2 to V4 and V6 to V8, the subject will consume successively the pastries which will have been assigned to him randomly and according to the randomization list.
  During the visit : A venous catheter will be placed by a medical biology technician and a blood sample will be taken immediately after placement: this is the first sample at T = 0 min. Then, the subject will have a maximum of 10 minutes to consume 294.1 g of elderflower madeleine (contained 50 g of glucose). The technician will then take blood samples at T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 minutes.
  Arms: a elderflower madeleine

SUMMARY:
In the early 1980s and following the first publications by Jenkins et al., The notion of glycemic index (GI) appeared with the aim of classifying the different sources of carbohydrates in our diet according to their effect on the post-prandial glycemic response. Since these years, many studies have been designed to determine the usefulness of the glycemic index and indicate that a low glycemic index for a food, a dish, a meal or a diet is associated with a decreased risk of metabolic pathologies (diabetes, hypertriglyceridemia), degenerative (cardiovascular diseases) or overload (obesity). This justifies the interest in favoring foods with a low glycemic index in healthy subjects.

A review confirmed the mechanistic link between postprandial blood sugar and the variability of blood sugar, making it possible, on the one hand, to maintain good glucose homeostasis and, on the other hand, to prevent pathologies such as obesity, diabetes and cardio-vascular diseases. The EFSA also considers that reducing the increase in blood sugar in the post-meal phase can be considered a physiological benefit, especially in subjects with glucose intolerance.

Post-meal blood sugar depends on many factors including the glycemic index of foods eaten during the meal. Knowing the glycemic index of foods is therefore very useful.

Mademoiselle Dessert offers pastries with a low glycemic index. The objective of this study is thus to determine the glycemic index of 6 pastries in order to inform consumers on these pastries glycemic index.

DETAILED DESCRIPTION:
The study will be carried out on healthy volunteers, aged from 18 to 65 with a body mass index (BMI) between 18 and 30 kg/m² (limits included).

The main objective of the study is to determine the glycemic index of 6 pastries in healthy volunteers with 7 kinetic points (0, 15, 30, 45, 60, 90 and 120 min).

ELIGIBILITY:
Inclusion Criteria:

* Man or woman ;
* Aged 18 to 65 (limits included);
* Having a body mass index (BMI) between 18 and 30 kg / m² (limits included);
* Agreeing to maintain their lifestyle (sport and diet) for the duration of the study;
* Agreeing not to smoke on the morning of each visit (before and during the visit).

Exclusion Criteria:

* Fasting blood glucose ≥ 6.1 mmol / L (or 1.10 g / L);
* Fasting triglycerides ˃ 2 g / L;
* Hyperinsulinemia (20 mIU / L) or history of insulinoma;
* Elevation of transaminases beyond 2x the upper limit;
* Subject presenting episodes of functional post-meal hypoglycaemia;
* Diabetic subject whether or not treated;
* Subject suffering from a severe eating disorder (anorexia, bulimia, binge eating);
* Subject presenting an immunodeficiency or any other serious pathology (cancer, hemopathy);
* Subject with a history of hypercholesterolemia and high blood pressure;
* Subject with renal failure;
* Subject with an allergy / intolerance to one of the constituents of the products under study;
* Subject with an intestinal pathology likely to modify digestion or absorption (Crohn's disease, etc.);
* Subject consuming more than 3 glasses of alcohol per day for men and more than 2 glasses per day for women;
* Subject not having a stable weight for the last 3 months (± 5%);
* Woman pregnant or planning to be during the study period, breastfeeding woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Glycemia: 7-point kinetics | 0 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 15 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 30 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 45 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 60 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 90 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8
Glycemia: 7-point kinetics | 120 min
  Blood glucose kinetics over 2 hours, performed from 7 blood samples and at 7 different times: T = 0, T = 15, T = 30, T = 45, T = 60, T = 90 and T = 120 min, on each test product and on the reference product (glucose).
  Visits V1 to V8

SECONDARY OUTCOMES:
Peak blood sugar (Cmax-Gly) | 0, 15, 30, 45, 60, 90 and 120 min
  For each product and from the glycemia and insulinemia dosage curves: peak blood sugar (Cmax-Gly).
  Visits V1 to V8
The time to onset of the blood sugar peak (Tmax-Gly) | 0, 15, 30, 45, 60, 90 and 120 min
  For each product and from the glycemia and insulinemia dosage curves: the time to onset of the blood sugar peak (Tmax-Gly). Visits V1 to V8
Insulin index | 0, 15, 30, 45, 60, 90 and 120 min
  For each product and from the glycemia and insulinemia dosage curves: insulin index Visits V1 to V8
Peak insulinemia (Cmax-Ins) | 0, 15, 30, 45, 60, 90 and 120 min
  For each product and from the glycemia and insulinemia dosage curves: peak insulinemia (Cmax-Ins).
  Visits V1 to V8
The time to onset of peak insulinemia (Tmax-Ins) | 0, 15, 30, 45, 60, 90 and 120 min
  For each product and from the glycemia and insulinemia dosage curves: the time to onset of peak insulinemia (Tmax-Ins). Visits V1 to V8

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel LECERF, MD, Principal Investigator — Institut Pasteur de Lille - NutrInvest
Locations (1):
- NutrInvest - Institut Pasteur de Lille, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: Undecided